CLINICAL TRIAL: NCT05758935
Title: Feasibility and Pilot Study of a Rule-based Chatbot Application for Adolescents With Anxiety Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 259293
Record Dates: First submitted 2023-01-17; First posted 2023-03-08 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Anxiety
Keywords: Adolescents; Anxiety; Chatbot intervention; Technology-delivered intervention
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mobile application (Experimental): A six weeks, rule-based chatbot intervention
  Interventions: Other: Rule-based chatbot intervention with therapist-guidance

INTERVENTIONS:
Other: Rule-based chatbot intervention with therapist-guidance — The intervention is a mobile application designed as a rule-based chatbot. The chatbot will present psychoeducational text, videos and ask questions based on cognitive behavioral techniques. The adolescents will receive weekly therapist support within the mobile application, in addition to weekly contact by phone. The intervention has a duration of six weeks, with a total of six modules.

SUMMARY:
The goal of this feasibility and pilot study is to investigate the feasibility and preliminary clinical effects of a new rule-based chatbot intervention for adolescents with anxiety symptoms. The main questions are:

* Is the intervention feasible for adolescents who are experiencing anxiety symptoms?
* How do the adolescents experience the use of the intervention?
* Does the intervention lead to a reduction in anxiety symptoms?
* Does the intervention lead to a clinically significant reliable improvement at functional level?

DETAILED DESCRIPTION:
Anxiety is one of the most common psychiatric disorders and the anxiety symptoms typically onsets in adolescence. The anxiety symptoms may be persistent into adulthood, leading to a poorer life quality and function impairments. The goal is to prevent the development of anxiety and comorbid disorders, as well as function impairment due to anxiety symptoms. This study wishes to investigate the feasibility and preliminary clinical effects of a digital intervention in an open pre-post and 3 months follow up study. The intervention consists of a rule-based click-chatbot, combined with therapist-guidance. This study will recruit N = 30 adolescents from Norway from age 13 up to 16 years old to investigate the feasibility and preliminary clinical effects of a rule-based click chatbot-intervention, and whether it causes a reduction in anxiety symptoms and increases of life functioning. If the intervention is feasible with promising results, the study will serve as a first step to a future randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* reporting anxiety symptoms that hinders them in participating in daily activities
* spending time trying to avoid these anxiety symptoms
* aged 13 and up to 16 years
* can read Norwegian

Exclusion Criteria:

* clinical cut-off on OCD subscale on RCADS-47> 10,
* clinical cut-off on Depression subscale on RCADS-47 > 16,
* ongoing treatment
* extensive reading/writing difficulties
* extensive concentration problems

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Revised Child Anxiety and Depression Scale -47 - Self-report | assessing change from screening, pre, immediately after the intervention, follow-up 1 month, and at follow-up 3 months
  anxiety and depressive symptoms, higher score indicates worse outcomes
Revised Child Anxiety and Depression Scale - 25 - Self-report | assessing change from week 2, and week 4
  short version of RCADS-47, measuring anxiety and depressive symptoms, with a higher score indicating worse symptoms
Revised Child Anxiety and Depression Scale -47 - Parent version | assessing change from pre, immediately after the intervention, follow-up 1 month, and at follow-up 3 months
  parent-reported anxiety and depressive symptoms, higher score indicates worse outcomes
Revised Child Anxiety and Depression Scale - 25 - Parent version | assessing change from week 2, and week 4
  parent-reported, short version of RCADS-47, measuring anxiety and depressive symptoms, with a higher score indicating worse symptoms

SECONDARY OUTCOMES:
Strengths and Difficulties Questionnaire - Youth version | assessing change from pre, immediately after the intervention, follow up 1 month, and at follow-up 3 months
  The scale measure adolescent's general mental health, with a higher score indicating worse symptoms. The study intends to use all three components of the measurement, including 1) the basis of SDQ, which includes 25 items on psychological attributes, 2) impact supplement, measuring functional level. The follow-up version also includes two additional follow-up questions
Strengths and Difficulties Questionnaire - Parent version | assessing change from pre, immediately after the intervention, follow up 1 month, and at follow-up 3 months
  The scale measure parent-reported adolescent's general mental health, with a higher score indicating worse symptoms. The study intends to use all three components of the measurement, including 1) the basis of SDQ, which includes 25 items on psychological attributes, 2) impact supplement, measuring the adolescents' functional level. The last component is used at follow up which also includes two additional follow-up questions

OTHER OUTCOMES:
Motivation Questionnaire | week 2
  assessments of their motivation to participate in the intervention, developed specifically for this study
Evaluation Questionnaire | immediately after the intervention
  evaluation assessments of the intervention, developed specifically for this study.
Demographics | pre-intervention
  gender, age

CONTACTS AND LOCATIONS:
Overall Officials: Smiti Kahlon, PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Research centre for digital mental health services, Haukeland University Hospital, Bergen, Vestland, Norway

IPD SHARING:
Plan to Share IPD: Yes
The full protocol and informed consent forms are available upon request. The datasets and the statistical code will not be publicly available, but may be available upon reasonable request through correspondence with principal investigator and according to the Norwegian law and regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: starting six months after publication
Access Criteria: IPD will be made available from PI on reasonable request and according to relevant Norwegian laws and regulations